CLINICAL TRIAL: NCT02770066
Title: A Prospective Danish National Registry of Percutaneous Transluminal Renal Angioplasty in Patients With Renovascular Hypertension
Brief Title: A Prospective Danish National Registry of PTRA in Patients With Renovascular Hypertension
Acronym: DAN-PTRA
Status: Recruiting | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Mark Reinhard, MD, PhD, University of Aarhus
Other Study IDs: DAN-PTRA
Record Dates: First submitted 2016-05-09; First posted 2016-05-12 (Estimated); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Renal Artery Obstruction; Hypertension, Renovascular; Cardiovascular Diseases; Kidney Diseases
MeSH Terms: conditions — Renal Artery Obstruction; Hypertension, Renovascular; Cardiovascular Diseases; Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Percutaneous transluminal renal angioplasty — Angioplasty plus stenting (angioplasty in patients with fibromuscular dysplasia)
  Adjuvant therapy in atherosclerotic renal artery stenosis - at the discretion of the treating physician
  * Antiplatelet therapy (usually standard)
  * Cholesterol-lowering drugs (usually standard)
  * Antihypertensive treatment with angiotensin-converting-enzyme inhibitor or angiotensin-receptor blocker (normally not contraindicated)
  * Smoking cessation, diet and physical activity (usually standard)

SUMMARY:
A prospective Danish national registry of percutaneous transluminal renal angioplasty (PTRA) in high-risk patients with renal artery stenosis selected on the basis of common national criteria, and with a common follow-up protocol for all three Danish centres offering PTRA

ELIGIBILITY:
Eligibility criteria

1. True resistant hypertension (≥ 3 antihypertensive drugs including a diuretic, if tolerated, and each prescribed at optimal doses) and uncontrolled blood pressure confirmed by 24-hour ambulatory blood pressure monitoring. The 24-hour ambulatory blood pressure monitoring is performed after nurse-administered medication and blood pressure measurements are performed hourly. If the average 24-hour ambulatory systolic blood pressure is ≥ 130 mmHg the patient can be evaluated for renal artery stenosis.
2. Hypertension and intolerance or side effects of the antihypertensive treatment. Hypertension is confirmed by 24-hour ambulatory blood pressure monitoring. The 24-hour ambulatory blood pressure monitoring is performed after nurse-administered medication and blood pressure measurements are performed hourly. If the average 24-hour ambulatory systolic blood pressure is ≥ 130 mmHg the patient can be evaluated for renal artery stenosis.
3. Progressive renal insufficiency (a reduction in eGFR > 5 ml/min/1,73 m2 per year) in patients with bilateral renal artery stenosis or in patients with renal artery stenosis and only one kidney.
4. Recurrent heart failure/pulmonary edema and resistant hypertension (≥ 3 antihypertensive drugs including a diuretic, if tolerated, and each prescribed at optimal doses) that may not be attributed to non-compliance, reduced left heart ventricular ejection fraction/heart valve disease or other obvious explanations (atrial fibrillation, fever, hyperthyroidism etc.). If the average 24-hour ambulatory systolic blood pressure is ≥ 130 mmHg after nurse-administered medication the patient can be evaluated for renal artery stenosis.
5. Younger patients (< 40 years) with hypertension (24-hour ambulatory blood pressure monitoring ≥ 130/80 mmHg after nurse-administered medication )

Inclusion Criteria:

All of the following:

1. At least one of the above eligibility criteria
2. Duplex doppler ultrasonography or renography investigations consistent with hemodynamically significant renal artery stenosis
3. CT angiography or renal arteriography with angiographic renal artery stenosis of ≥ 70 % reduction of the luminal diameter in at least one projection

Exclusion Criteria:

1. If angiography/arteriography, ultrasonography or renography is consistent with bilateral significant renal artery stenosis and only one side is treated with PTRA
2. PTRA of a renal artery supplying a kidney which pre-PTRA handles ≤ 10% of the total kidney function (with no blockage of the renin-angiotensin system) and has a kidney size < 7 cm (length)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: High-risk patients with renal artery stenosis
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2015-01-01; Primary Completion 2030-01 (Estimated); Study Completion 2035-01 (Estimated)

PRIMARY OUTCOMES:
Changes in 24-hour ambulatory systolic and diastolic blood pressures from baseline to 24 months after PTRA in patients with 24-hour ambulatory average systolic blood pressure ≥ 150 mmHg at baseline | Measured 24 months post-PTRA
  Changes in 24-hour ambulatory systolic and diastolic blood pressures (calculated from hourly means) from baseline to 24 months after percutaneous transluminal renal angioplasty in patients with 24-hour ambulatory average systolic blood pressure ≥ 150 mmHg at baseline and with significant artery stenosis either
  1. Unilaterally (one or two kidneys)
  2. Bilaterally with treatment of both kidneys
  All 24-hour ambulatory blood pressure measurements are performed after nurse-administered medication. Likewise, it will below be inferred that renal artery stenosis is defined as in the primary endpoint.

SECONDARY OUTCOMES:
Changes in 24-hour ambulatory systolic and diastolic blood pressures from baseline to 24 months after PTRA in patients with 24-hour ambulatory average systolic blood pressure ≥ 130 mmHg at baseline | Measured 24 months post-PTRA
  Changes in 24-hour ambulatory systolic and diastolic blood pressures (calculated from hourly means) from baseline to 24 months after percutaneous transluminal renal angioplasty in patients with 24-hour ambulatory average systolic blood pressure ≥ 130 mmHg at baseline and with significant artery stenosis
Changes in 24-hour ambulatory systolic and diastolic blood pressures (statistically adjusted for treatment changes) from baseline to 24 months after PTRA in patients with 24-hour ambulatory average systolic blood pressure ≥ 150 mmHg at baseline | Measured 24 months post-PTRA
  Changes in 24-hour ambulatory systolic and diastolic blood pressures (calculated from hourly means) (statistically adjusted for treatment changes) from baseline to 24 months after percutaneous transluminal renal angioplasty in patients with 24-hour ambulatory average systolic blood pressure ≥ 150 mmHg at baseline and with significant artery stenosis
Changes in 24-hour ambulatory systolic and diastolic blood pressures (statistically adjusted for treatment changes) from baseline to 24 months after PTRA in patients with 24-hour ambulatory average systolic blood pressure ≥ 130 mmHg at baseline | Measured 24 months post-PTRA
  Changes in 24-hour ambulatory systolic and diastolic blood pressures (calculated from hourly means) (statistically adjusted for treatment changes) from baseline to 24 months after percutaneous transluminal renal angioplasty in patients with 24-hour ambulatory average systolic blood pressure ≥ 130 mmHg at baseline and with significant artery stenosis
Changes in 24-hour ambulatory systolic and diastolic blood pressures (unadjusted and statistically adjusted for treatment changes) | Measured at 3, 12, 36, 48 and 60 months
  Changes in 24-hour ambulatory systolic and diastolic blood pressures (unadjusted and statistically adjusted for treatment changes) from baseline to 3, 12, 36, 48 and 60 months after PTRA in patients with 24-hour ambulatory average systolic blood pressure ≥ 150 mmHg and in patients with 24-hour ambulatory average systolic blood pressure ≥ 130 mmHg
Change in antihypertensive treatment (defined daily doses) | Measured at 3, 12, 24, 36, 48 and 60 months
Change in kidney function | Measured at 3, 12, 24, 36, 48 and 60 months
  Change in estimated glomerular filtration rate (eGFR) and change in percentage side distribution measured by renography at baseline and 24 months after PTRA
Clinical composite end point | Measured at 3, 12, 24, 36, 48 and 60 months
  Clinical composite end point
  1. death from cardiovascular causes
  2. death from renal causes
  3. stroke
  4. myocardial infarction
  5. hospitalization for congestive heart failure
  6. progressive renal insufficiency (a reduction from baseline of 30% or more in eGFR)
  7. permanent renal-replacement therapy
  Only the first event per participant is included in the composite
Safety composite end point (< 30 days after PTRA) | Measured at 3, 12, 24, 36, 48 and 60 months
  Safety composite end point (< 30 days after PTRA)
  1. all cause mortality
  2. rupture, dissection, perforation or occlusion of renal artery
  3. critical bleeding (need of blood transfusion)
  4. embolization
  5. significant loss of kidney function (reduction from baseline of 30% or more in eGFR)
  6. ipsilateral nephrectomy
  7. pseudoaneurysm formation
  8. stent thrombosis
  Only the first event per participant is included in the composite

CONTACTS AND LOCATIONS:
Locations (5):
- Denmark (5):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus N
  - Glostrup University Hospital/ Rigshospitalet, Glostrup Municipality
  - Holbaek Hospital, Holbæk
  - Odense University Hospital, Odense C

REFERENCES:
- [Derived] Reinhard M, Schousboe K, Andersen UB, Buus NH, Rantanen JM, Bech JN, Mafi HM, Langfeldt S, Bharadwaz A, Horlyck A, Jensen MK, Jeppesen J, Olsen MH, Jacobsen IA, Bibby BM, Christensen KL. Renal Artery Stenting in Consecutive High-Risk Patients With Atherosclerotic Renovascular Disease: A Prospective 2-Center Cohort Study. J Am Heart Assoc. 2022 Apr 5;11(7):e024421. doi: 10.1161/JAHA.121.024421. Epub 2022 Mar 24. PMID 35322677